CLINICAL TRIAL: NCT06684262
Title: Comparison of the Effect of Erector Spina Plane Block and Intraperitoneal Local Anesthetic Infiltration on the Quality of Postoperative Recovery in Patients Undergoing Laparoscopic Cholecystectomy.
Brief Title: Intraperitoneal Local Anesthetic Infiltration Versus Erector Spinae Block in Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hakan Duzla MD, Research Assistant, Ankara University
Other Study IDs: 2024000006-4
Record Dates: First submitted 2024-04-01; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Quality of Recovery; Postoperative Analgesia
Keywords: Erector Spina Plane Block; intraperitoneal instillation of local anesthetics; Postoperative quality of recovery; Postoperative analgesia; laparoscopic cholecystectomy; intraperitoneal infiltration of local anaesthetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group IPLA: Following the extraction of the gallbladder, the surgical team promptly administers a 45 mL local anesthetic solution blend consisting of 20 mL of bupivacaine at a concentration of 0.5%, 10 mL of lidocaine at a concentration of 2%, and 15 mL of 0.9% saline solution to the gallbladder bed and subdiaphragmatic region. This administration is performed via an aspiration catheter under direct visualization provided by the laparoscopic camera
- Group ESP: At the end of the operation and before tracheal extubation, patients will be turned into the lateral decubitus position. Bilateral erector spinae plane block will be applied at the T8 spinous process level. Under asepsis-antisepsis standards, a 12 mHz linear ultrasound probe will be placed approximately 3 cm lateral to the spinous process of the T8 vertebra in a longitudinal parasagittal orientation. After identification of the trapezius, rhomboid major, erector spinae muscles and transverse process, an aspiration test using an 80 mm peripheral nerve block needle, 22.5 ml of local anesthetic mixture (10 mL bupivacaine at 0.5% concentration, 5 mL lidocaine at 2% concentration, 7.5 mL 0.9% NaCl) will be applied bilaterally.

SUMMARY:
Laparoscopic cholecystectomy is a commonly performed intra-abdominal surgical procedure all over the world. It may take an average of 4-5 weeks for patients to return to their pre-operative quality of life and standards after this surgery. Both Erector Spinae Plane Block and Intraperitoneal Local Anesthetic Infiltration method are methods used to reduce postoperative pain. However, there is no study in the literature comparing these 2 methods in terms of postoperative recovery quality. In this study, patients will receive Erector Spinae Plane Block or Intraperitoneal Local Anesthetic Infiltration at the end of surgery, and both techniques will be compared using the preoperative and postoperative quality of recovery 40 survey.

DETAILED DESCRIPTION:
The Preoperative Quality of Recovery 40 questionnaire will be administered to patients scheduled for laparoscopic cholecystectomy who consent to participate in the study. Following the surgical procedure, patients will receive either intraperitoneal local anesthetic infiltration or bilateral erector spinae plane block for postoperative analgesia. These interventions will be examined in an observational study comprising two distinct groups. At the 24-hour mark postoperatively, the Quality of Recovery 40 (QoR 40) survey will be readministered to the patients, and the outcomes will be subjected to comparative analysis. Throughout the postoperative period, patients in both cohorts will be closely monitored. Pain scores and opioid-associated adverse effects (such as nausea, vomiting, and pruritus) will be assessed at the 1st, 2nd, 4th, 8th, 12th, and 24th hours. Subsequent to the surgical procedure, patients in both groups will be provided with morphine via patient-controlled analgesia, and the extent of opioid consumption within the first 24 hours postoperatively will be compared.

Primary purpose: To compare the effects of Erector Spina Plane (ESP) block and intraperitoneal local anesthetic infiltration on the quality of postoperative recovery in patients undergoing laparoscopic cholecystectomy.

Secondary objectives: To compare the effects of ESP block and intraperitoneal local anesthetic infiltration on postoperative pain scores at rest and with movement, total opioid consumption, and incidence of opioid-related side effects in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Will undergo laparoscopic cholecystectomy operation,
* Patients with an American Society of Anesthesiologists Physical Status Score (ASA-PS) of 1, 2 and 3 will be included.

Exclusion Criteria:

* Patients who do not give consent
* Those who are allergic to the drugs used in the research
* Those with coagulation disorders
* Having a history of alcohol and substance use
* Having a history of serious psychiatric and neurological diseases
* Having chronic pain syndrome
* Those with local infection in the area to be blocked
* Patients with sepsis and undergoing emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Will undergo laparoscopic cholecystectomy operation,
  * Patients with an American Society of Anesthesiologists Physical Status Score (ASA-PS) of 1, 2 and 3 will be included.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Quality of postoperative recovery | postoperative 24th hour
  The aim of this study was to use the Quality of Recovery 40 questionnaire as a method to evaluate and compare the effects of Erector Spinae Plane (ESP) block and intraperitoneal local anesthetic infiltration on the quality of postoperative recovery in patients undergoing laparoscopic cholecystectomy. The QoR-40 questionnaire is a self-assessment questionnaire used to evaluate the quality of postoperative recovery. It is a questionnaire that evaluates the level of pain, physical and emotional status of patients and consists of 40 questions and five domains: emotional status (n=9), comfort (n=12), psychological support (n=7), physical independence (n=5) and pain (n=7). Each question is scored on a 5-point Likert scale ranging from 1 to 5. The total score ranges from 40 (worst quality of recovery) to 200 (best quality of recovery). A low total score indicates poor quality of recovery; a high total score indicates good quality of recovery.

SECONDARY OUTCOMES:
Postoperative pain | Postoperative 1st-2nd-4th-8th-12th-24th hours
  To evaluate and contrast the impact of Erector Spinae Plane (ESP) block and intraperitoneal local anesthetic infiltration on postoperative pain levels during rest and movement, as measured by the numerical pain rating scale (ranging from 0 to 10, with 0 representing no pain and 10 representing the worst possible pain), among patients undergoing laparoscopic cholecystectomy.Higher numerical pain scale scores indicate higher pain levels, and lower scores indicate lower pain levels.
Postoperative opioid consumption | for 24 hours postoperatively
  To compare the 24-hour postoperative morphine consumption in milligrams after Erector Spinae Plane (ESP) block and intraperitoneal local anesthetic infiltration.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided